CLINICAL TRIAL: NCT00052611
Title: Celecoxib In Biomarker Modulation Of Oral Precancerous Lesions: A Pilot Study
Brief Title: Celecoxib in Preventing Cancer in Patients With Oral Leukoplakia and/or Head and Neck Dysplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lori J. Wirth, MD, Wirth, Lori MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-024; P30CA006516 (NIH); DFCI-02024; DFCI-2002-P-00150/2
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Head and Neck Cancer
Keywords: lip and oral cavity cancer; paranasal sinus and nasal cavity cancer; hypopharyngeal cancer; laryngeal cancer; oropharyngeal cancer; nasopharyngeal cancer; salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Oropharyngeal Neoplasms; Nasopharyngeal Neoplasms; Salivary Gland Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Celecoxib (Experimental): Celecoxib will be given at a pre-determine dose twice daily for 3 months. If there is a favorable change in biomarker expression on biopsy at 3 months, treatment will continue to complete a 12-month treatment period.
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib
  Other Names: Celebrex

SUMMARY:
Patient at increased risk for developing a new head and neck squamous cell carcinoma are invited to take part in this study.

The investigators of this trial will attempt to study the effectiveness of Celecoxib in preventing cancer in patients who have oral leukoplakia and/or head and neck dysplasia.

DETAILED DESCRIPTION:
Celecoxib is being studied in precancerous lesions of the head and neck in part because, it has been shown to prevent the progression of another type of precancerous polyps (a type of abnormal growth) in patients at high risk for colorectal cancer. There are, however, no published studies yet looking at this drug in humans for the prevention of head and neck cancers. The U.S. Food and Drug Administration has approved celecoxib for arthritis and the prevention of polyps in patients with familial adenomatous polyposis (a type of precancerous syndrome in some families that can lead to colon cancer).

This study is being done to find out several things:

* Is celecoxib, also known by the trade name Celebrex ®, effective in reducing the expression of precancerous markers (biological signals for specific cellular activities) in oral leukoplakia and dysplasia (abnormal growth) of the oral mucosa?
* Is celecoxib effective in reducing the size of oral leukoplalda lesions and/or presence of dysplasia?
* Does the reduction in precancerous markers correspond with reduction of oral leukoplalda and/or presence of dysplasia?
* What are the side effects of celecoxib in this patient population?

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be ≥ 18 years.
* Subjects will have oral leukoplakia on clinical examination and/or more than one previous HNSCC with dysplasia histologically proven on random biopsy within 6 months at the time of entry.
* Patients who have had surgical treatment for a previous HNSCC, stage I-III, will be eligible for enrollment if they are cancer-free ≥ 9 months at the time of entry. Patients with CIS or new leukoplakia will be immediately eligible if they are more then 9 months from treatment of a prior carcinoma.
* Leukoplakia lesions must be ≥ 0.5 cm in at least one dimension to be considered measurable. Measurable lesions are not required for entry.
* The ECOG performance status will be ≤ 2. (See Appendix B for ECOG performance status.)
* The life expectancy will be ≥12 months.
* Subjects will have adequate organ function with a platelet count of >100,000, ANC > 1500, PT and PTT < 1.5 X ULN, creatinine <1.5, urine protein <2+, and total bilirubin and liver transaminases <1.5 X ULN.
* Premenopausal women will be required to use a reliable method of birth control throughout the course of therapy.
* Subjects will provide written, voluntary informed consent

Exclusion Criteria:

* Patients who have had surgical treatment for a previous HNSCC, stage I-III, will not be eligible for enrollment if they are cancer-free < 9 months at the time of entry.
* Subjects with contraindication to nasopharyngoscopy and biopsy will not be enrolled.
* Significant comorbidities, including known coronary artery disease, angina, history of myocardial infarction, congestive heart failure of at least grade 2 according to the New York Heart Association Criteria, advanced COPD requiring use of home oxygen, active alcohol abuse, bleeding diathesis, any history of gastrointestinal ulcer, acute or chronic renal insufficiency, or acute or chronic liver disease, will preclude enrollment in the trial.
* Enrollment in the trial will be limited to patients who are free from current tobacco use. If the patient has a history of previous tobacco use, they Must be abstinent for at least 1 month prior to enrollment and meet the criteria established by the Food and Drug Administration for assessing smoking cessation, i.e. have not taken even a puff or taste of tobacco, including cigarette, cigar, pipe, chewing tobacco or other tobacco products, in the past 4 weeks.
* Any active malignancy, except non-melanoma skin cancer, will preclude enrollment.
* Persons who have taken full-dose aspirin, NSAIDs, COX-2 inhibitors and systemicallyabsorbed steroids, including inhaled steroids and nasal steroids other than mometazone, at least 3 times per week for 2 or more consecutive weeks within 3 months of enrollment will be excluded. Persons who have taken retinoids or selenium within 3 months of enrollment, or who have a history of anaphylactoid reaction to aspirin, NSAIDs or COX- 2 inhibitors will not be enrolled.
* Persons taking ACE inhibitors will not be enrolled. Diuretics for CHF, or treatment with lithium or fluconazole will also preclude enrollment. Patients on coumadin will be required to have PT/INR monitoring BIW after starting celecoxib, until the patient is on a stable dose of coumadin for 7 days, and must have no contraindication to holding the coumadin for study biopsies.
* Pregnant, lactating women or premenopausal women with a positive f3HCG will not be enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2002-06 (Actual); Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Response Rate Of PGE2 | 2 years

SECONDARY OUTCOMES:
Change In SEB Expression Of COX-2 | 2 years
Response Of Measurable Lesions | 2 years
Assessing Safety | 2 years
Change In SEB Expression Of Akt | 2 years
Change In SEB Expression Of Ki-67 | 2 years
Change In SEB Expression Of BCL2 | 2 years
Change In SEB Expression Of BAX | 2 years
Change In SEB Expression Of VEGF | 2 years
Change In SEB Expression Of CD31 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lori J. Wirth, MD, Study Chair — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No